CLINICAL TRIAL: NCT05819164
Title: Comparison of Multiple Oxygenation Targets With Different Oximeters in COPD and Non-COPD Patients- Impact on Oxygen Flows
Brief Title: Comparison of Multiple Oxygenation Targets With Different Oximeters in Chronic Obstructive Pulmonary Disease (COPD) and Non-COPD Patients- Impact on Oxygen Flows
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, Principal Investigator, Laval University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-4002
Record Dates: First submitted 2023-04-03; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: COPD Exacerbation; Pneumonia; Hypoxemia; Respiratory Disease
Keywords: oxygen, oximeter
MeSH Terms: conditions — Pneumonia; Hypoxia; Respiration Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 88% SpO2 target (Experimental): During this periods , oxygen will be administered in manual titration to reach 88% of SpO2.
  Interventions: Device: Masimo oximeter; Device: Nellcor oximeter; Device: Nonin oximeter
- 90% SpO2 target (Experimental): During this periods , oxygen will be administered in manual titration to reach 90% of SpO2.
  Interventions: Device: Masimo oximeter; Device: Nellcor oximeter; Device: Nonin oximeter
- 92% SpO2 target (Experimental): During this periods , oxygen will be administered in manual titration to reach 92% of SpO2.
  Interventions: Device: Masimo oximeter; Device: Nellcor oximeter; Device: Nonin oximeter
- 94% SpO2 target (Experimental): During this periods , oxygen will be administered in manual titration to reach 94% of SpO2.
  Interventions: Device: Masimo oximeter; Device: Nellcor oximeter; Device: Nonin oximeter
- 96% SpO2 target (Experimental): During this periods , oxygen will be administered in manual titration to reach 96% of SpO2.
  Interventions: Device: Masimo oximeter; Device: Nellcor oximeter; Device: Nonin oximeter

INTERVENTIONS:
Device: Masimo oximeter — During this period, the Masimo oximeter Radical 7 was used for SpO2 reading
Device: Nellcor oximeter — During this period, the Nellcor oximeter N-600 was used for SpO2 reading
Device: Nonin oximeter — During this period, the Nonin oximeter was used for SpO2 reading

SUMMARY:
The oximeter is an instrument for monitoring patients receiving oxygen therapy. It displays pulse oxygen saturation (SpO2), which is a reflection of arterial oxygen saturation (SaO2). An accurate SpO2 value is essential for optimal management of the O2 flow delivered to patients. Several factors can influence this measurement and the choice of ventilatory support: the type of oximeter used, skin pigmentation and the oxygenation goal.

The objective of our study is to evaluate the impact of the oxygenation goal and the oximeter used on oxygen flows in patients with COPD (or with hypercapnia, or at risk of hypercapnia) and in patients without COPD (in particular pneumonia, pulmonary fibrosis and other pathologies) Our hypothesis is that the SpO2 target and oximeter used will have an impact on oxygen flows and that these effects will be synergistic in these different populations.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* On conventional oxygen therapy with SpO2 between 88 and 100% with the usual oximeter and nasal cannula.
* SpO2 < 92% in ambient air with the usual oximeter

Exclusion Criteria:

* No availability of the SpO2 signal with the usual oximeter
* False nails or nail polish
* Severe anemia documented on the last blood count during the current hospitalization (Hb < 80g/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-22 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxygen flow | assessed up to 10 minutes
  the mean oxygen flow to reach the SpO2 target +/- 1% during 2 minutes for each period and each oximeter

SECONDARY OUTCOMES:
Partial oxygen weaning | assessed up to 10 minutes - until SpO2 target stability for 2 minutes
  Rate of partial oxygen weaning (Oxygen flow <=0.5 L/min) to reach the SpO2 target for each period and each oximeter
Complete oxygen weaning | assessed up to 10 minutes - until SpO2 target stability for 2 minutes
  Rate of complete oxygen weaning (Oxygen flow <=0.1 L/min) to reach the SpO2 target for each period and each oximeter
High oxygen flow | assessed up to 10 minutes - until SpO2 target stability for 2 minutes
  Rate of high oxygen flow (Oxygen flow >5.0 L/min) to reach the SpO2 target for each period and each oximeter
Oximeter bias comparison | assessed up to 10 minutes - until SpO2 target stability for 2 minutes
  the mean bias between the result of the different oximeter

IPD SHARING:
Plan to Share IPD: No